CLINICAL TRIAL: NCT01284205
Title: Randomized, Double-blind, Multi-center Study Comparing MCC to BCG as First Line Immunotherapy in Patients With Non-muscle Invasive (Superficial) Bladder Cancer at High Risk of Recurrence or Progression
Brief Title: First Line Comparative Study of EN3348 (MCC) vs BCG in NMIBC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This indication is not being pursued at this point in time.
Sponsor: Bioniche Life Sciences Inc. (Industry)
Responsible Party: Director of CRND, Endo Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EN3348-302
Expanded Access: Available
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Bladder Cancer
Keywords: non-muscle invasive bladder cancer; superficial bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCC (Experimental): Intravesical Administration of Mycobacterial Cell-Wall DNA Complex
  Interventions: Biological: Mycobacterial Cell-Wall DNA Complex
- BCG (Active Comparator): Intravesical Administration of Bacillus Calmette-Guerin
  Interventions: Biological: Bacillus Calmette-Guerin

INTERVENTIONS:
Biological: Mycobacterial Cell-Wall DNA Complex — 8 mg/50 mL (sterile WFI) Intravesical Administration; one weekly instillation per week for 6 week Induction Phase; three weekly instillations per month at Months 3, 6, 12, 18, and 24 followed by Maintenance Phase.
  Arms: MCC
Biological: Bacillus Calmette-Guerin — mg/50 mL (sterile saline) Intravesical Administration; one weekly instillation per week for 6 week Induction Phase; three weekly instillations per month at Months 3, 6, 12, 18, and 24 followed by Maintenance Phase.
  Arms: BCG

SUMMARY:
The purpose of this study is to compare the safety and efficacy of EN3348 (MCC) versus BCG as first line treatment in patients with non-muscle invasive bladder cancer that are at high risk for recurrence or progression.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed urothelial carcinoma of the bladder (high grade Ta or T1 papillary lesions, CIS)
* histologically confirmed diagnosis within 42 days of study treatment
* life expectancy of greater than 5 years
* ECOG performance status of 2 or less
* absence of urothelial carcinoma involving the upper urinary tract or prostatic urethra within 12 months from start of study treatment

Exclusion Criteria:

* current or previous history of muscle invasive bladder tumors (>T2)
* current or previous history of lymph node and/or distant metastases from bladder cancer
* current evidence of squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the bladder
* current systemic cancer therapy
* previous immunotherapy for bladder cancer
* previous intravesical chemotherapy treatment
* contraindication to use BCG of known tolerance to BCG
* history of malignancy of any organ system within the past 5 years (with the exception of basal cell or squamous cell carcinoma, stage T1 prostate cancer, carcinoma in situ of the cervix, colon polyps)
* patients who cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy or biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Duration of disease-free survival (time to recurrence, progression or death) in all patients | Baseline, Month 3, 6, 9, 12, 15, 18, 21, and 24
Percent of patients who due to study drug-related AEs experience 2 consecutive treatment delays or discontinue due to drug related AEs | Baseline through 24 months

SECONDARY OUTCOMES:
Disease-free survival rate at 2 years | Month 24
Frequency, severity, and nature of drug-related AEs | Baseline through 24 Months
Duration of progression-free survival (time to progression or death) in all patients | Baseline, Month 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48 and 60
Frequency, severity, and nature of drug-related SAEs | Baseline through 24 months
Number of treatment delays and their reason | Baseline, Month 3, 6, 9, 12, 15, 18, 21, and 24
Frequency, severity and nature of all AEs | Baseline through 24 months
Number of treatment discontinuations and their reason | Baseline through 24 months
Duration of Survival (time to death from any cause) in all patients | Baseline through month 60

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Laguna Hills, California
  - Los Angeles, California
  - San Diego, California
  - Englewood, Colorado
  - Daytona Beach, Florida
  - Overland Park, Kansas
  - Shreveport, Louisiana
  - Garden City, New York
  - New York, New York
  - Pittsburgh, Pennsylvania
  - Myrtle Beach, South Carolina
  - McAllen, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia